CLINICAL TRIAL: NCT03568474
Title: Postoperative Pain After Application of Silver Diamine Fluoride and Glass Ionomer Versus Glass Ionomer Alone Following Minimal Caries Removal Technique in Asymptomatic Young Permanent Teeth With Deep Caries. A Randomized Pilot Study.
Brief Title: Silver Diamine Fluoride After Minimal Caries Removal Technique in Asymptomatic Young Permanent Teeth With Deep Caries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehan Anwar Ibrahim, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Egypt Cairo University
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Deep Caries
MeSH Terms: interventions — silver diamine fluoride; glass ionomer

STUDY DESIGN:
Intervention Model Description: parallel two arm groups with 1:1 allocation ratio
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant, care provider, outcomes assessor and statistician will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Silver Diamine Fluoride (Experimental): Silver Diamine fluoride will be applied after after minimal caries removal then glass ionomer over it followed by composite resin restoration.
  Interventions: Drug: Silver Diamine Fluoride; Drug: Glass Ionomer
- Glass Ionomer (Active Comparator): Glass ionomer will be applied after minimal caries removal followed by composite resin restoration.
  Interventions: Drug: Glass Ionomer

INTERVENTIONS:
Drug: Silver Diamine Fluoride — Indirect pulp capping material
  Other Names: SDF
  Arms: Silver Diamine Fluoride
Drug: Glass Ionomer — Indirect pulp capping material
  Other Names: GI

SUMMARY:
This study is comparing between the Silver Diamine Fluoride after minimal caries removal versus glass ionomer in permanent teeth with open apex

DETAILED DESCRIPTION:
The study will be carried on young permanent molars with open apices & with deep caries. Incomplete caries removal and application of indirect pulp capping materials where Silver Diamine Fluoride (Group I) will be compared with glass ionomer only (group II). Then final restoration with composite resin for both groups. Children will be followed up for 9 months.

ELIGIBILITY:
Inclusion criteria:

1. Patients free from any systematic diseases.
2. Young permanent molars with incompletely formed roots having deep carious lesions according to clinical and radiographic examination and at risk of pulp exposure if complete caries is removed.
3. Absence of clinical pathologic signs (fistula, swelling and abnormal tooth mobility)
4. The absence of clinical symptoms of irreversible pulpitis.
5. Absence of adverse radiographic findings (interradicular or periapical radiolucencies, thickening of the periodontal space, internal and external root resorption).
6. Compliant patient/ parent.

Exclusion criteria:

1. Teeth with previous restorative treatment.
2. Unrestorable teeth.
3. Uncooperative patients.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 9 months
  Will be assessed by questioning the patient or the guardian whether there is postoperative pain or not, Binary (yes or no)

SECONDARY OUTCOMES:
Tooth vitality | 9 months
  Will be assessed by Vitality test using thermal stimulation, binary (yes or no)
Abscess | 9 months
  Will be assessed intraoral Clinical examination whether there is swelling or not, binary (yes or no)
Pain on percussion | 9 months
  Will be assessed by Percussion test by using the back of the mirror on the tooth, binary (yes or no)
Root lengthening | 9 months
  Will be assessed measuring the root length by mm on the digital radiography (digora software)

CONTACTS AND LOCATIONS:
Overall Officials: Nevine G Waly, Professor, Study Chair — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Sara A Mahmoud, PhD, Study Director — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Mohamed K Zayt, PhD, Study Director — Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University; Rehan A Ibrahim, MSc, Principal Investigator — Pediatric Dentistry, Faculty of Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: Yes
thesis and article publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after cessation of the study
Access Criteria: Internet